CLINICAL TRIAL: NCT05827796
Title: A Phase Ib/II, Open-label Clinical Study to Evaluate the Safety, Tolerability and Antitumor Activities of IN10018+Standard Chemotherapy and IN10018+Standard Chemotherapy+KN046 in Subjects With Advanced Pancreatic Cancer
Brief Title: IN10018+ Standard Chemotherapy (+KN046) in Subjects With Advanced Pancreatic Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: InxMed (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IN10018-012
Record Dates: First submitted 2023-03-28; First posted 2023-04-25 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Albumin-Bound Paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1: IN10018+ standard chemotherapy (albumin-bound paclitaxel + gemcitabine) (Experimental): Subjects will be treated with IN10018 25 mg/50 mg/100 mg, once daily, oral+ albumin-bound paclitaxel 125 mg/m2 IV infusion on Days 1 and 8 of each 21-Day Cycle+ gemcitabine 1000 mg/m2 IV infusion on Days 1 and 8 of each 21-Day Cycle.
  Interventions: Drug: IN10018; Drug: Albumin-Bound Paclitaxel; Drug: Gemcitabine
- Cohort 2: IN10018+ standard chemotherapy (albumin-bound paclitaxel + gemcitabine)+KN046 (Experimental): Subjects will be treated with IN10018 25 mg/50 mg/100 mg, once daily, oral+ albumin-bound paclitaxel 125 mg/m2 IV infusion on Days 2 and 8 of each 21-Day Cycle+ gemcitabine 1000 mg/m2 IV infusion on Days 2 and 9 of each 21-Day Cycle+KN046 5 mg/kg IV infusion on Day 1 of each 21-Day Cycle.
  Interventions: Drug: IN10018; Drug: Albumin-Bound Paclitaxel; Drug: Gemcitabine; Drug: KN046

INTERVENTIONS:
Drug: IN10018 — IN10018 orally once daily at approximately the same time each day, to ensure a dosing interval of approximately 24 hours.
  Other Names: BI853520
Drug: Albumin-Bound Paclitaxel — Albumin-bound paclitaxel will be administered as per the schedule specified in the respective arm.
Drug: Gemcitabine — Gemcitabine will be administered as per the schedule specified in the respective arm.
Drug: KN046 — KN046 5 mg/kg on Day 1 of each 21-Day Cycle.
  Arms: Cohort 2: IN10018+ standard chemotherapy (albumin-bound paclitaxel + gemcitabine)+KN046

SUMMARY:
This study is a multicenter, open-label, single-arm, phase Ib/II clinical study comprising two phases: dose confirmation phase and dose expansion phase. The objective of the dose confirmation phase is to determine the recommended Phase II dose (RP2D) of IN10018+ standard chemotherapy (albumin-bound paclitaxel + gemcitabine) and IN10018 + KN046 + standard chemotherapy in subjects with advanced pancreatic cancer. The dose expansion phase will further explore the antitumor activities and safety of combination therapy in subjects with advanced pancreatic cancer.

DETAILED DESCRIPTION:
This is a multicenter, open-label, single-arm, phase Ib/II clinical study to evaluate the safety, tolerability, and antitumor activities of IN10018 + standard chemotherapy (albumin paclitaxel + gemcitabine) and IN10018 + KN046 + standard chemotherapy in subjects with advanced pancreatic cancer.

This study includes two cohorts, Cohort 1: IN10018 + standard chemotherapy; Cohort 2: IN10018 + standard chemotherapy + KN046. Each cohort consists of 2 phases: a dose confirmation phase and a dose expansion phase. The dose confirmation phase aims to determine recommended Phase II dose (RP2D) of IN10018+ standard chemotherapy and IN10018 + KN046 + standard chemotherapy in subjects with advanced pancreatic cancer. The dose expansion phase will further explore the antitumor activities and safety of combination therapy in subjects with advanced pancreatic cancer.

According to the Package Insert of standard chemotherapy (albumin paclitaxel and gemcitabine), the Investigator's Brochure (IB) and drug characteristics of KN046, it is expected that IN10018 has little possibility of interaction with standard chemotherapy and KN046, and the safety characteristics are clearly non-overlapping. The therapeutic dose of KN046, albumin-bound paclitaxel and gemcitabine are fixed in this study. In the dose confirmation phase, IN10018 dose will be modified according to the causality between dose-limiting toxicities (DLTs) and IN10018.

ELIGIBILITY:
Inclusion Criteria:

1. With a full understanding of the study, each subject voluntarily agreed to participate in this study and sign the informed consent form.
2. Female or male subjects ≥ 18 years at the time of signing informed consent.
3. Histological or cytology-confirmed pancreatic ductal adenocarcinoma (including adenosquamous carcinoma).
4. No previous systemic treatment for unresectable, locally advanced, or metastatic pancreatic cancer.
5. At least one measurable lesion per RECIST 1.1.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
7. Life expectancy of at least 3 months as assessed by the investigator.
8. Must have recovered from all AEs due to previous anticancer therapies to ≤ Grade 1 (CTCAE 5.0) or stable status as assessed by the investigator. Subjects with any grade of alopecia and grade 2 peripheral neuropathy could be enrolled.
9. Adequate bone marrow, liver, renal, and coagulation function .
10. A female subject is eligible to participate if she is not pregnant, not breastfeeding, and at least 1 of the following conditions applies:

    * Not a woman of childbearing potential (WOCBP) . or
    * A WOCBP who agrees to follow the contraceptive guidance.

Exclusion Criteria:

1. Has had major surgery or major trauma within 28 days prior to the first dose of study treatment.
2. Has known BRCA1/2 mutations.
3. Has received prior systemic anticancer therapy including chemotherapy, targeted therapy, immunotherapy, unmarketed investigational drugs or therapy within 28 days prior to the first dose of study treatment.
4. Previous anti-programmed death 1(PD-1), anti-programmed death-ligand 1 (PD-L1), or anti-cytotoxic T lymphocyte-associated antigen-4 (CTLA-4) antibody therapy, or any other antibody or drug that specifically targets T-cell co-stimulation or checkpoint pathways, or prior treatment with focal adhesion kinase (FAK) inhibitors.
5. Has received radical radiotherapy within 3 months prior to the first dose of study treatment. Subjects who have received palliative radiotherapy with a local standardized dose within 2 weeks prior to the first dose of study treatment.
6. Has received previous allogeneic hematopoietic stem cell transplantation or organ transplantation.
7. Has received live vaccines and live attenuated vaccines within 28 days prior to the first dose of study treatment.
8. Has interstitial pneumonia or lung disease.
9. History or current active autoimmune diseases.
10. Has a prior history of other malignancy, other than cured cutaneous squamous cell carcinoma, basal cell cancer, non-basal invasive bladder cancer, and prostate/cervical/breast cancer in situ within 5 years prior to the first dose of study treatment.
11. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
12. Has a history of major cardiovascular, cerebrovascular or thromboembolic diseases within 6 months before the first dose of study treatment.
13. Active infection with poor systemic treatment control.
14. Has known human immunodeficiency virus (HIV) infection, active hepatitis B virus (HBV) or hepatitis C (HCV) infection, or active syphilis and tuberculosis.
15. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-12-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Related Adverse Events （AEs） | 1 year
  Incidence and severity of AEs, with severity determined according to the NationalCancer Institute Common Terminology Criteria for Adverse Events, Version 5.0 (NCI CTCAE v5.0)
To evaluate the objective response rate (ORR) per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) in subjects with advanced pancreatic cancer. | 2 years
  Proportion of subjects who have the best objective response of either complete response (CR) or partial response (PR), as assessed by the investigator.

SECONDARY OUTCOMES:
Disease Control Rate (DCR) per RECIST 1.1, as evaluated by investigators | 1 year
  Proportion of subjects who have CR, PR, or stable disease (SD).
duration of response (DoR) per RECIST 1.1, as evaluated by investigators | 1 years
  Available for subjects who demonstrate CR or PR, DoR is defined as the time from the first evidence of CR or PR until progressive disease (PD) or death due to any cause, whichever occurs first, as assessed by the investigator.
Progression free survival (PFS) per RECIST 1.1, as evaluated by investigators | 1 years
  Defined as the time from the first day of study treatment to the first disease progression or death due to any cause, whichever occurs first.
Overall survival (OS) | 2 years
  Defined as the time from the first day of study treatment to death due to any cause.
Incidence of Treatment-Related AEs | 2 years
  Incidence and severity of AEs, with severity determined according to the NCI CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Liwei Wang, Principal Investigator — Renji Hospital of Shanghai Jiaotong University of Medicine
Locations (1):
- Renji Hospital of Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No